CLINICAL TRIAL: NCT04764786
Title: Polyphenol Enriched Extra-virgin Olive Oil and Postprandial Glucose Response in Patients With Type 1 Diabetes: Possible Effects and Mechanisms
Brief Title: Polyphenol Enriched Extra-virgin Olive Oil and Postprandial Glycemia in Type 1 Diabetes (DOP)
Acronym: DOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 37/19
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; postprandial glycemia; polyphenols
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVOO+POLY (Experimental): Acute test meal
  Interventions: Other: EVOO+POLY
- OO-POLY (Active Comparator): Acute test meal
  Interventions: Other: OO-POLY

INTERVENTIONS:
Other: EVOO+POLY — a test meal seasoned with extra virgin olive oil rich in polyphenols
  Arms: EVOO+POLY
Other: OO-POLY — a test meal seasoned with olive oil poor in polyphenols
  Arms: OO-POLY

SUMMARY:
The aims of this study are to investigate the short term effects of MUFA alone vs. MUFA plus Polyphenols contained in the extra-virgin olive oil (EVOO) on the postprandial glycemic response in patients with type 1 diabetes and to explore the possible mechanisms through which MUFA alone or MUFA plus Polyphenols contained in EVOO could influence postprandial glycaemia.The intervention will be preceded by two-weeks run-in period during which participants will consume an usual olive oil, fill-in a 7-day dietary food record and practice continuous blood glucose monitoring (CGM) in order to optimize basal insulin infusion values and the insulin-to-glycemic load ratio.The study will be conducted according to a randomized cross-over design.

The participants will consume, in random order at a distance of one week from each other, a meal-test seasoned with extra virgin olive oil rich in polyphenols (EVOO + POLY) or a meal-test seasoned with olive oil poor in polyphenols (OO-POLY). Upon fasting and during the 6 hours following the meal, patients will undergo to:

1. Venous blood drawing samples for the evaluation of gastrointestinal hormones, markers of systemic inflammation and oxidative stress.
2. Breath test with 13C-octanoic acid, for the study of gastric emptying. During the experimental period the participants will undergo to continuous glucose monitoring wearing sensors 7 days/week.

The results of this study will allow optimizing insulin therapy based on the macronutrient composition of the meal in patients with type 1 diabetes mellitus treated with insulin pump. This will improve glycemic control and quality of life of these patients and reduce the risk of developing chronic diabetes complications.

DETAILED DESCRIPTION:
In a recent study the use of extra virgin olive oil (EVOO) (rich in MUFA) to a high glycemic index meal attenuated the early PGR observed when this meal were consumed with either low-fat or butter (rich in SAFA), while low glycemic index foods determined a blunted early postprandial response and a late rise of blood glucose levels, independently of type and quantity of fat added. Of relevance, the effects on PGR of dietary components known to influence postprandial blood glucose metabolism, such as polyphenols, remain completely unexplored in patients with T1D. Polyphenols are bioactive compounds with high antioxidant power highly present also in EVOO, which could have contributed to the favorable effects on PGR that the investigators observed in patients with T1D.

The aims of this study are to investigate the short term effects of MUFA alone vs. MUFA plus Polyphenols contained in EVOO on the postprandial glycemic response in patients with type 1 diabetes and to explore the possible mechanisms through which MUFA alone or MUFA plus Polyphenols contained in EVOO could influence postprandial glycaemia.

Patients with type 1 diabetes treated with continuous subcutaneous insulin infusion for at least 6 months and HbA1c less than 8.5%, will be recruited at the diabetes care unit of the Federico II University teaching hospital.

The intervention will be preceded by two-weeks run-in period during which participants will consume an usual olive oil, fill-in a 7-day dietary food record and practice continuous blood glucose monitoring (CGM) in order to optimize basal insulin infusion values and the insulin-to-glycemic load ratio.The study will be conducted according to a randomized cross-over design.

The participants will consume, in random order at a distance of one week from each other, a meal-test seasoned with extra virgin olive oil rich in polyphenols (EVOO + POLY), or a meal-test seasoned with olive oil poor in polyphenols (OO- POLY). Upon fasting and during the 6 hours following the meal, patients will undergo to:

1. Venous blood drawing samples for the evaluation of gastrointestinal hormones, markers of systemic inflammation and oxidative stress.
2. Breath test with 13C-octanoic acid, for the study of gastric emptying. During the experimental period the participants will undergo to continuous glucose monitoring wearing their sensors 7 days/week.

The meals will be similar in terms of glycemic load and macronutrient composition and will differ in the type of seasoning used.

The test meal will be postponed in case of premeal blood glucose levels outside the 90-150 mg/dl range or a rapid decrease/increase of glucose levels (above 1 mg/dl per min) during the previous 60 min according to CGM measurement, Pre-meal insulin doses, will be calculated based on the individual insulin-to-glycemic load ratio and will be the same on all two occasions.

At the end of the experimental period, data from CGM and insulin pump will be downloaded by dedicated informatics platforms. Participants will use the CGM system integrated with the insulin pump, i.e., the one they are accustomed to.

The primary outcome will be the difference between the postprandial blood glucose change groups following dietary interventions and it will be evaluated by 2-way ANOVA for repeated measurements.

The results of this study will allow optimizing insulin therapy based on the macronutrient composition of the meal in patients with type 1 diabetes mellitus treated with insulin pump. This will improve glycemic control and quality of life of these patients and reduce the risk of developing chronic diabetes complications. These complications involve severe disability for patients and huge costs for the community.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with continuous subcutaneous insulin infusion for at least 6 months
* HbA1c less than 8.5% (69 mmol/mol)

Exclusion Criteria:

* Pregnancy and breastfeeding
* Any other chronic or acute disease apart diabetes seriously affecting health status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
the between-group difference in postprandial glycemia changes after the dietary interventions | 6 hours
  Postprandial incremental area (iAUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Napoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No